CLINICAL TRIAL: NCT03189381
Title: A Pilot Phase 2 Study Evaluating Dose De-escalation in Whole Brain Radiation Therapy With Simultaneous Integrated Boost for Patients With Brain Metastases
Brief Title: Pilot Phase 2 Study Whole Brain Radiation Therapy With Simultaneous Integrated Boost for Patients With Brain Metastases
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early termination leading to no patients enrolled in cohort B.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kevin Shiue, MD, Assistant Professor, Indiana University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IUSCC-0605
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Results first posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Brain Metastases
Keywords: Whole Brain Radiation; Simultaneous Integrated Boost
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Cohort A (Experimental): Standard PCI dose
  Interventions: Radiation: Cohort A
- Cohort B (Experimental): Low PCI dose
  Interventions: Radiation: Cohort B

INTERVENTIONS:
Radiation: Cohort A — Cohort A - WBRT dose = 25 Gy, SIB dose = 42 Gy, # of daily fractions = 10, SIB dose in EQD2 = 49.7 Gy
  Arms: Cohort A
Radiation: Cohort B — Cohort B - WBRT dose = 20 Gy, SIB dose = 40 Gy, # of daily fractions = 8, SIB dose in EQD2 = 50.0 Gy
  Arms: Cohort B

SUMMARY:
This trial is a pilot, Phase 2, sequential two-cohort study designed to test two de-escalated whole brain radiation therapy (WBRT) dose levels and assess their ability to maintain acceptable in-brain distant control. The WBRT dose would decrease as the study moves forward, both in terms of absolute value and equivalent dose in 2 Gray fractions (EQD2) (as determined by the linear quadratic radiobiological model). The absolute value of the simultaneous integrated boost (SIB) dose will change with each dose level because the number of fractions delivered will depend on the WBRT dose. As such, the SIB dose will be manipulated such that the EQD2 will remain essentially equivalent despite the difference in the number of fractions delivered. This design will ensure that the only variable is the change in WBRT dose.

The concept is that WBRT with SIB would be expected to maximize both local and in-brain distant control as has already been shown in studies exploring WBRT with SRS boost. However, by itself WBRT with SIB does not address the concern over neurocognitive outcomes. Therefore, investigators hypothesize that there is a lower WBRT dose threshold that will maintain acceptable in-brain distant control, particularly in the setting of a SIB to gross lesions to maintain treated lesion control. In addition, lower overall brain dose (including lower hippocampal dose without specific hippocampal avoidance) may potentially improve neurocognitive function. Investigators are also interested in evaluating treated lesion control, overall survival, neurocognitive sequelae of therapy, quality of life, performance status, and adverse effects of therapy. Biomarker identification for potential correlative circulating tumor DNA and microRNA is an exploratory endpoint to generate data for future prospective evaluation.

DETAILED DESCRIPTION:
Primary Objective Evaluate two de-escalated whole brain radiation dose levels (in the setting of simultaneous integrated boost to gross lesions) with respect to in-brain distant control for brain metastases, defined as an in-brain failure rate outside of the planning target volume at 6 months of < 20%.

Secondary Objectives

1. Evaluate treated lesion control at 6 months for brain metastases in the setting of a predetermined total biologically effective SIB dose as determined by radiographic progression within the planning target volume with fusion and overlay of follow-up MRIs.
2. Evaluate overall survival at 6 months for brain metastases in the setting of WBRT with SIB.
3. Evaluate changes in neurocognitive function after WBRT with SIB in the following domains: verbal learning and memory as assessed by the Hopkins Verbal Learning Test - Revised (HVLT-R).
4. Evaluate changes in health-related quality of life as assessed by the Functional Assessment of Cancer Therapy with Brain Subscale (FACT-Br) after WBRT-SIB for brain metastases.
5. Evaluate changes in performance status as assessed by the Karnofsky Performance Status tool after WBRT-SIB for brain metastases.
6. Evaluate adverse events after WBRT-SIB for brain metastases according to current CTCAE criteria.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 at time of consent.
2. Ability to provide written informed consent and HIPAA authorization.
3. Pathological diagnosis of any solid tumor histology (from any site in the body).
4. Pathological or clinical (i.e., by imaging) diagnosis of brain metastatic tumor lesions.
5. Total volume of lesions ≤ 30 cm3.
6. Maximum volume of largest lesion ≤ 5 cm3.

   a. This volume limit would be equivalent to a largest diameter of about 2.1 cm, assuming a perfect sphere.
7. Not a candidate for or eligible for but refused Gamma Knife radiosurgery.

Exclusion Criteria

1. Previous radiation to the brain, including WBRT or brain radiosurgery.
2. Life expectancy < 6 months (as estimated per current ds-GPA).
3. For histologies not included in the ds-GPA publications or otherwise noted online at brainmetgpa.com, the PI will use either published or validated data, or the PI's best clinical judgment to determine the patient's expected survival.
4. Inability to comply with treatment per investigator discretion.
5. Inability to complete neurocognitive assessments per investigator discretion.

Of note, tumor lesion number is not an inclusion or exclusion criteria as we are using volume-based criteria instead.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin R. Shiue, MD, Principal Investigator — Indiana University School of Medicine
Locations (3):
- United States (3):
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Methodist Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Standard prophylactic intracranial irradiation (PCI) dose
  Cohort A: whole-brain radiation therapy dose (WBRT) = 25 Gy, simultaneous integrated boost (SIB) dose = 42 Gy, # of daily fractions = 10, SIB dose in equivalent dose in 2 Gray fractions (EQD2) = 49.7 Gy
- Cohort B: Low prophylactic intracranial irradiation (PCI) dose
  Cohort B: Cohort B - whole-brain radiation therapy dose (WBRT) dose = 20 Gy, simultaneous integrated boost (SIB) dose = 40 Gy, # of daily fractions = 8, SIB dose in equivalent dose in 2 Gray fractions (EQD2) = 50.0 Gy
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 20 | 0
Completed | 19 | 0
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are given for patients who had a treatment start date and were deemed eligible.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 20 | 0 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (15.12) |  | 59.8 (15.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 |  | 11
  Male | 9 |  | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 19 |  | 19
  Unknown or Not Reported | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 3 |  | 3
  White | 17 |  | 17
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 |  | 20
Primary Cancer Diagnosis [Count of Participants; unit: Participants]
  Bladder | 1 |  | 1
  Breast | 5 |  | 5
  Colon | 1 |  | 1
  Kidney | 1 |  | 1
  Lung | 11 |  | 11
  Skin - Scalp and Neck | 1 |  | 1
Number of Lesions at Baseline [Median (Inter-Quartile Range); unit: lesions] | 7.00 [4.75 to 8.75] |  | 7.00 [4.75 to 8.75]
Number of Boosted Lesions at Baseline [Median (Inter-Quartile Range); unit: lesions] | 7.00 [4.00 to 8.25] |  | 7.00 [4.00 to 8.25]

OUTCOME MEASURES:

1. Primary Outcome: In-Brain Distant Failure Rate
Description: An actuarial 6-month rate of new parenchymal lesions seen outside the planning target volume of any lesion that received SIB on any post-treatment MRI (in all 3 planes). This is the binomial proportion of patients who experienced in-brain distant failure by 6 months and the associated 95% confidence interval.
Time Frame: 6 Months
Population: Includes the patients evaluable for in-brain distant failure at 6 months. There were no patients accrued in cohort B.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 9 | 0
proportion of patients | 0.444 [0.137 to 0.788] |

2. Secondary Outcome: Treated Lesion Local Control
Description: An actuarial 6-month rate of any new, recurrent, or progressing (as defined by Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria) tumor within the planning target volume on any post-treatment MRI. This details the estimated 6-month survival and associated 95% confidence interval from the Kaplan Meier method. The time from treatment start to local failure was calculated. Patients who did not experience local failure were censored at the date last know alive or at the date of death if they expired.
Time Frame: 6 Months
Population: Includes patients evaluable for 6-month outcomes. There were no patients accrued in cohort B.
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 9 | 0
survival probability | 1.000 [1.000 to 1.000] |

3. Secondary Outcome: Overall Survival for Evaluable Patients
Description: An actuarial 6-month rate of patients still alive regardless of disease status. This details the estimated 6-month survival and associated 95% confidence interval from the Kaplan Meier method. For patients who expired, the time from treatment start to death was calculated. Patients who did not expire were censored at the date last know alive.
Time Frame: 6 Months
Population: Includes patients evaluable for 6-month outcomes. There were no patients accrued in cohort B.
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 9 | 0
survival probability | 1.000 [1.000 to 1.000] |

4. Secondary Outcome: Change in Neurocognitive Function From Baseline to 6 Months
Description: The change in scores from the neurocognitive test were calculated by subtracting the baseline score from the 6-month score. Positive values indicate an increase from baseline and negative values indicate a decrease.
  The neurological test scores were assessed with the Hopkins Verbal Learning Test - Revised (HVLT). In the HVLT, 12 nouns are read and the participant is asked to recall in 3 rounds. Total words recalled are summed for the Total Recall score ranging from 0-36 (higher score represents better recall). The delayed recall score is tested 20-25 mins after the initial recall and ranges from 0-12 (higher scores are better). Retention (%) is the percentage of words recalled and ranges from 0-100 (higher values represent better recall). The recognition discrimination score is tested by a series of yes/no responses from the participant identifying 12 words from a list of 24 and subtracts the number of true positives minus the true negatives (higher values are better).
Time Frame: 6 Months
Population: Includes patients evaluable for 6-month outcomes. There were no patients accrued in cohort B.
Measure: Median (Inter-Quartile Range); unit: difference in score on a scale
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 9 | 0
difference in score on a scale
  Total Recall Raw Score | -1.00 [-2.25 to 0.25] |
  Delayed Recall Raw Score | -1.00 [-2.75 to 0.25] |
  Recognition Discrimination Index Raw Score | 0.00 [-2.75 to 0.00] |

5. Secondary Outcome: Change in Health-Related Quality of Life (QoL) From Baseline to 6 Months
Description: The change in scores of health-related quality of life test from baseline to 6 months calculated by subtracting the baseline score from the 6-month score. Positive values indicate an increase in score from baseline to 6 months while negative values indicate a decrease.
  The Functional Assessment of Cancer Therapy with Brain Subscale (FACT-Br) asks questions on a scale from 0 to 4 with 0 being "not at all" and 4 being "very much". Responses were reversed, if applicable, and compiled to calculate physical well-being (range: 0-28), social/family well-being (range: 0-28), emotional well-being (range: 0-24), functional well-being (range: 0-28), bone marrow transplant (BMT) (range: 0-40), and brain cancer (range: 0-92) subscale scores. These subscale scores were then summed to obtain the trail outcome index (range: 0-148), bone marrow transplant (FACT-BMT) (range: 0-96), general (FACT-G) (range: 0-108), and FACT-Br (range: 0-200) total scores. The higher the score, the better the QoL.
Time Frame: 6 Months
Population: Includes patients evaluable for 6-month outcomes. There were no patients accrued in cohort B.
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 9 | 0
scores on a scale
  Physical Well-Being | -1.00 [-2.00 to 1.00] |
  Social/Family Well-Being | -2.00 [-2.00 to 1.00] |
  Emotional Well-Being | -1.00 [-2.00 to 0.00] |
  Functional Well-Being | -1.00 [-3.00 to 1.00] |
  Bone Marrow Transplant (BMT) Subscale | 0.00 [-3.00 to 2.00] |
  Trial Outcome Index | -4.00 [-6.00 to 1.00] |
  FACT-G | -2.00 [-7.00 to 4.00] |
  FACT-BMT | -1.00 [-8.00 to 3.83] |

6. Secondary Outcome: Change in Performance Status
Description: Total change in performance status score was calculated by substracting the baseline score from the follow-up score. Positive values indicate an increase in score from baseline while negative values indicate a decrease in score from baseline. Functional status evaluated using the Karnofsky Performance Score (KPS) Index. The KPS score is evaluated on a scale from 0 to 100 where 0 is death and 100 is "normal no complaints; no evidence of disease".
Time Frame: 12 Months
Population: Includes patients evaluable for 6-month outcomes. There were no patients accrued in cohort B.
Measure: Median (Inter-Quartile Range); unit: difference in score on a scale
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 9 | 0
difference in score on a scale
  Baseline to 3 Months | -10.00 [-10.00 to 10.00] |
  Baseline to 6 Months | 0.00 [0.00 to 0.00] |
  Baseline to 12 Months | 0.00 [0.00 to 5.00] |

7. Secondary Outcome: Incidence of Early and Late Treatment-Related Adverse Effects
Description: This is the percentage of eligible patients who experienced the respective treatment-related AE while on study. Adverse effects (AEs) were defined per CTCAE and considered treatment-related if the AE start date occurred on or after the first date of treatment and it was possibly, probably, or definitely related to treatment. AEs were recorded from the start of treatment until the patient was off-study.
Time Frame: Up To 39 Months
Population: Includes the patients marked as eligible who started treatment. There were no patients accrued in cohort B.
Measure: Number; unit: percentage of patients
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 20 | 0
percentage of patients
  Fatigue | 50.00 |
  Alopecia | 30.00 |
  Memory Impairment | 25.00 |
  Headache | 10.00 |
  Somnolence | 10.00 |
  Blurred Vision | 5.00 |
  Cognitive Disturbance | 5.00 |
  Dermatitis Radiation | 5.00 |
  Dry Skin | 5.00 |
  Mucosal Infection | 5.00 |
  Oral Pain | 5.00 |
  Papulopustular Rash | 5.00 |
  Pruritus | 5.00 |
  Rash Maculo-Papular | 5.00 |
  Skin and Subcutaneous Tissue Disorders | 5.00 |
  Vomiting | 5.00 |

8. Secondary Outcome: Overall Survival for Eligible Patients
Description: as for outcome 3
Time Frame: 6 Months
Population: Includes patients who started treatment and were deemed eligible for the study. There were no patients accrued in cohort B.
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 20 | 0
survival probability | 0.700 [0.451 to 0.853] |

9. Secondary Outcome: Change in Neurocognitive Function Retention Percentage Raw Score From Baseline to 6 Months
Description: as for outcome 4
Time Frame: 6 Months
Population: Includes patients evaluable for 6-month outcomes. There were no patients accrued in cohort B.
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 9 | 0
percentage | -3.00 [-30.50 to 2.25] |

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study and assessed up to 39 months
Description: There were no patients accrued in cohort B. Therefore, the number at risk for all events is zero.
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 15/20 | 0/0
Serious Adverse Events (participants affected / at risk) | 9/20 | 0/0
Other Adverse Events (participants affected / at risk) | 20/20 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=20) | Cohort B (N=0)
Abdominal pain (Gastrointestinal disorders) | 1 | NA
Breast infection (Infections and infestations) | 1 | NA
Confusion (Psychiatric disorders) | 1 | NA
Dehydration (Metabolism and nutrition disorders) | 1 | NA
Dysarthria (Nervous system disorders) | 1 | NA
Dysphagia (Gastrointestinal disorders) | 1 | NA
Encephalopathy (Nervous system disorders) | 1 | NA
Fall (Injury, poisoning and procedural complications) | 1 | NA
Gait disturbance (General disorders) | 1 | NA
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | NA
Hallucinations (Psychiatric disorders) | 1 | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Neutrophil count decreased (Investigations) | 1 | NA
Sepsis (Infections and infestations) | 1 | NA
Thromboembolic event (Vascular disorders) | 1 | NA
Urinary tract infection (Infections and infestations) | 1 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=20) | Cohort B (N=0)
Fatigue (General disorders) | 13 | NA
Headache (Nervous system disorders) | 7 | NA
Alopecia (Skin and subcutaneous tissue disorders) | 6 | NA
Nausea (Gastrointestinal disorders) | 6 | NA
Anorexia (Metabolism and nutrition disorders) | 5 | NA
Edema limbs (General disorders) | 5 | NA
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 | NA
Memory impairment (Nervous system disorders) | 5 | NA
Vomiting (Gastrointestinal disorders) | 5 | NA
Abdominal pain (Gastrointestinal disorders) | 4 | NA
Blurred vision (Eye disorders) | 4 | NA
Constipation (Gastrointestinal disorders) | 4 | NA
Diarrhea (Gastrointestinal disorders) | 4 | NA
Dysphagia (Gastrointestinal disorders) | 4 | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | NA
Somnolence (Nervous system disorders) | 4 | NA
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 | NA
Anxiety (Psychiatric disorders) | 3 | NA
Dysgeusia (Nervous system disorders) | 3 | NA
Fall (Injury, poisoning and procedural complications) | 3 | NA
Mucosal infection (Infections and infestations) | 3 | NA
Thromboembolic event (Vascular disorders) | 3 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | NA
Ataxia (Nervous system disorders) | 2 | NA
Bruising (Injury, poisoning and procedural complications) | 2 | NA
Chills (General disorders) | 2 | NA
Confusion (Psychiatric disorders) | 2 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | NA
Dehydration (Metabolism and nutrition disorders) | 2 | NA
Dizziness (Nervous system disorders) | 2 | NA
Fever (General disorders) | 2 | NA
Gait disturbance (General disorders) | 2 | NA
Hypoglycemia (Metabolism and nutrition disorders) | 2 | NA
Infections and infestations - Other, specify (Infections and infestations) | 2 | NA
Insomnia (Psychiatric disorders) | 2 | NA
Leukocytosis (Blood and lymphatic system disorders) | 2 | NA
Lymphocyte count decreased (Investigations) | 2 | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | NA
Oral pain (Gastrointestinal disorders) | 2 | NA
Papulopustular rash (Infections and infestations) | 2 | NA
Peripheral motor neuropathy (Nervous system disorders) | 2 | NA
Pruritus (Skin and subcutaneous tissue disorders) | 2 | NA
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 | NA
Urinary tract infection (Infections and infestations) | 2 | NA
Weight loss (Investigations) | 2 | NA
Anemia (Blood and lymphatic system disorders) | 1 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 | NA
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 | NA
Breast infection (Infections and infestations) | 1 | NA
Cardiac troponin I increased (Investigations) | 1 | NA
Chest pain - cardiac (Cardiac disorders) | 1 | NA
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | NA
Cognitive disturbance (Nervous system disorders) | 1 | NA
Depressed level of consciousness (Nervous system disorders) | 1 | NA
Depression (Psychiatric disorders) | 1 | NA
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | NA
Dry mouth (Gastrointestinal disorders) | 1 | NA
Dry skin (Skin and subcutaneous tissue disorders) | 1 | NA
Dysarthria (Nervous system disorders) | 1 | NA
Encephalopathy (Nervous system disorders) | 1 | NA
Esophageal pain (Gastrointestinal disorders) | 1 | NA
Fracture (Injury, poisoning and procedural complications) | 1 | NA
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | NA
Hallucinations (Psychiatric disorders) | 1 | NA
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | NA
Hypocalcemia (Metabolism and nutrition disorders) | 1 | NA
Hypokalemia (Metabolism and nutrition disorders) | 1 | NA
Hyponatremia (Metabolism and nutrition disorders) | 1 | NA
Hypotension (Vascular disorders) | 1 | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | NA
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | NA
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | NA
Neutrophil count decreased (Investigations) | 1 | NA
Pain (General disorders) | 1 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | NA
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | NA
Palpitations (Cardiac disorders) | 1 | NA
Pelvic pain (Reproductive system and breast disorders) | 1 | NA
Peripheral sensory neuropathy (Nervous system disorders) | 1 | NA
Platelet count decreased (Investigations) | 1 | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Portal vein thrombosis (Hepatobiliary disorders) | 1 | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | NA
Seizure (Nervous system disorders) | 1 | NA
Sepsis (Infections and infestations) | 1 | NA
Sinus tachycardia (Cardiac disorders) | 1 | NA
Tremor (Nervous system disorders) | 1 | NA
Urinary retention (Renal and urinary disorders) | 1 | NA
Ventricular tachycardia (Cardiac disorders) | 1 | NA
Watering eyes (Eye disorders) | 1 | NA
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | NA
White blood cell decreased (Investigations) | 1 | NA
Wound complication (Injury, poisoning and procedural complications) | 1 | NA

LIMITATIONS AND CAVEATS:
Early termination leading to no patients enrolled in cohort B.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT03189381/Prot_SAP_000.pdf